CLINICAL TRIAL: NCT04598100
Title: Promoting Resiliency in Veteran Families With Young Children
Acronym: FOCUS-EC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Patricia E. Lester, MD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: R01HD072324-05 (NIH)
Record Dates: First submitted 2020-10-01; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Stress, Psychological; Stress Disorders, Traumatic; Regulation, Self; Behavior, Child; Emotional Stress; Trauma, Psychological; Anxiety; Depression
Keywords: resilience; families; children; intervention; deployment
MeSH Terms: conditions — Stress, Psychological; Stress Disorders, Traumatic; Self-Control; Child Behavior; Psychological Trauma; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FOCUS-EC (Active Comparator): FOCUS-EC provides developmental guidance, parent education, and key resilience skills that promote positive individual and family coping, including emotional regulation, problem solving, goal setting, communication, and management of deployment & combat stress reminders, which foster parent-child and family cohesion. The intervention is delivered in six 90-minute sessions in the family home. Each session is structured with a check-in, review of the previous week's "home activity," primary activity and discussion, selection of a new "home activity", and a closing check-out. The family learns and practices the skills during the sessions, commits to practicing the skills during the week, and reports on their experiences the following session so that skills can be reinforced and adjustments made. FOCUS-EC promotes parenting skills and more cohesive family relationships in two key phases: 1) creating a family deployment and reintegration timeline and 2) enhancing parent-child interactions.
  Interventions: Behavioral: FOCUS-EC
- Web-Based Family Education (No Intervention): Families in the WB condition will be provided access to online educational materials covering topics such as typical child development, effects of early childhood separations, common child reactions to family stress, and the importance of self-care. CDM families in this condition will also have access to the standard services that are available to OEF/OIF/OND veterans through the VHA system, TriCare, and California Department of Veterans Affairs.

INTERVENTIONS:
Behavioral: FOCUS-EC
  Arms: FOCUS-EC

SUMMARY:
Family-centered prevention services for civilian dwelling military (CDM) families & children are rarely available in civilian communities or often framed around mental disorders and family deficits. As of June 2010, over 1 million military service members from various military conflicts have become veterans. Wartime deployments can adversely impact the psychological health of children as well as marital relationships, parent-child relationships & overall family functioning. Although young children in CDM families may never have to cope with another parental deployment, their families may continue to struggle with the lasting effects of wartime deployment that cannot be ameliorated by singularly treating the service member. There is a need for family-centered preventive interventions that effectively build resilience and mitigate war deployment-related family difficulties, especially given the potential adverse emotional & developmental impact of deployment separations and reintegration stress on young children and their parents. To address this need, this study proposes to test the efficacy of FOCUS-EC (Families OverComing Under Stress for Early Childhood), an established strength-based, family-centered preventive intervention that is culturally sensitive and socially accepted by active duty military communities & has promising program evaluation data. A randomized control trial will be conducted with 200 CDM families with young children, ages 3 to 5 years, recruited from Los Angeles & surrounding counties (200 veterans, 150 spouses, and 300 children). CDM families will be randomized to the FOCUS-EC intervention condition (n=100 families; 100 veterans, 75 spouses, 150 children) or web-based educational materials condition (n=100 families; 100 veterans, 75 spouses, and 150 children) and assessed at baseline, 3, 6, & 12 months. It is hypothesized that in the FOCUS-EC condition: 1) children will exhibit more positive social-emotional & behavioral outcomes & developmental competencies than children in the comparison condition, 2) families will exhibit more positive family environment, improved parenting, enhanced parent-child relationships, & fewer parent psychological health problems than families in the comparison condition. The investigators also aim to explore potential moderating effects of child health/development risk, military & deployment/separation history, exposure to combat/trauma during deployment, and veteran & spouse/partner background factors.

DETAILED DESCRIPTION:
In Phase I, the investigators modified FOCUS-EC for CDM families with young children, and developed a platform for the web-based educational materials. The intervention manual, training materials and assessments were also finalized. The research team already has well-developed manuals for FOCUS-EC, including an intervention manual, technical assistance manual, and training curriculum that have been used for various settings. Existing materials have been customized for CDM families and will be housed online. Materials will include information about child development and common reactions to early separations, as well as deployment and family stress. The team also has extensive experience developing online education for military families (for example, see www.focusproject.org). Online educational information is a common governmental strategy to serve CDM families; the proposed design enables a rigorous comparison of a facilitator-led interactive intervention (FOCUS-EC) to the provision of standardized online resources. Finally in Phase 1, to ensure that FOCUS-EC would meet the unique needs of CDM families, intervention sessions were modified and conducted with CDM families. The investigators believe that this customization with a small group of CMD families has been sufficient to identify the emerging needs of CDM families (e.g., challenges associated with the transition to civilian life, renegotiating family roles more permanently, shifting control or power between parents, reestablishing family routines and rituals, and redefining family relationships), incorporate culturally sensitive language that is common to this population, and tailor the FOCUS-EC for a home visit delivery model. Themes, current concerns, and language identified were incorporated into the FOCUS-EC for CDM families protocol. A similar approach was used to ensure that language used in FOCUS-EC was appropriate for various branches of the service in the preliminary work. The finalized intervention manual and training includes protocols and back-up procedures for clinical emergencies and ethical issues, as documented in the current technical assistance manual.

Phase 2:

All families will complete a baseline assessment, consisting of questionnaires, brief interviews, and family observational tasks.

After the baseline assessment, the family will be randomized into either the FOCUS-EC condition or a web-based education condition. Simple block randomization will be done. Families will be assigned to either the intervention or web-based resources control condition using a computer-generated randomization list with block sizes of 2, 4, and 6. The code for this randomization process can be found at: http://biostat.mc.vanderbilt.edu/wiki/Main/BlockRandomizationwithRandomBlockSizes. No stratification will be done for gender, age, site, etc.

Participants who are randomized to the web-based education condition will be provided with an account and password to a study-developed/supported website that will provide online resources with content comparable to and consistent with FOCUS-EC intervention sessions. That is, web-based materials will provide information on parent-child communication, emotion regulation, problem-solving, stress management, and family resilience. Participants will not be required to utilize these resources; they may access this website as often as they choose and implement the information and strategies as they wish.

These families will also complete the exact same assessments as those families in the intervention condition. In addition, they will answer a questionnaire assessing various aspects of the web-based resources (e.g., usefulness, ease of use/navigation, frequency of use, etc.).

Participants who are randomized to the FOCUS-EC condition will participate in six intervention sessions.

The FOCUS-EC protocols and measures have been finalized, programmed, and tested, and informed consent protocols were developed. FOCUS-EC will be delivered using a tele-health 6 session manualized protocol. Sessions will be led by trained, Master's level facilitators leading virtual home visiting sessions. FOCUS-EC is framed within a skill-building and relationship-strengthening psycho-educational model that integrates research on traumatic stress, child development, and the military-developed combat operational stress continuum model for prevention. FOCUS-EC provides developmental guidance, parent education, and key resilience skills that promote positive individual and family coping, including emotional regulation, problem solving, goal setting, communication, and management of deployment and combat stress reminders, which foster parent-child and family cohesion. The intervention is delivered in six 45-90-minute sessions in the family's home via a computer, internet connection, and webcam . Each session is structured with a check-in, review of the previous week's "home activity," primary activity and discussion, selection of a new "home activity" for the week, and a closing check-out. The family learns and practices the skills during the sessions, commits to practicing the skills during the week, and reports on their experiences the following session so that skills can be reinforced and any necessary adjustments can be made. FOCUS-EC promotes parenting skills and more cohesive family relationships in two key phases: 1) creating a family deployment timeline and 2) enhancing parent-child interactions (see figure 3). In the first phase, parents develop a family deployment narrative which fosters understanding, communication, mutual support, and positive co-parenting across the parenting dyad (session 1 and 2). This stage begins with a web-based family psychological health "check-in" utilizing innovative programming already established by this team, and utilized by families in service settings. This check-in serves to assist the facilitator and the family in identifying strengths and areas of concern in the initial session through use of standardized psychological health screening instruments (see Appendix). Parents set goals for what they are motivated to achieve during program participation. Parents also recount a narrative timeline for their deployment/separation and reintegration history. Through perspective taking and active listening, parents bridge estrangements and enhance their understanding of their child's reactions to deployments and separations, co-parenting, and family leadership. In the second phase, parents work on enhancing parent-child interactions in a series of parent-only education and parent-child practice sessions. In these alternating sessions, parents model and help their children with emotional identification and communication; learn and practice basic play, attunement, and relationship-enhancement strategies; increase awareness of trauma, loss, and separation reminders that impact effective parenting; practice behavior management techniques; elicit a developmentally appropriate narrative of their child's experiences; and plan for the future.

The study team has experience with a number of innovative technologies designed to deliver in-home preventive interventions utilizing a virtual delivery platform, including a secure in-home "teleprevention" platform. This platform has been implemented through a service delivery model pilot and has demonstrated the feasibility of remote/virtual home visits, including a video-teleconferencing platform which enables participants to access sessions using secure software (e.g., "Go To Meeting"). In home access to computers and internet in this population is high; thus, it anticipated that this will not be a barrier to enrollment and participation. All core intervention components and activities have been adapted for remote delivery platform modifications, intervention training, delivery and technical support manuals.

ELIGIBILITY:
Inclusion Criteria:

* • Non-active duty OEF/OIF/OND veteran with at least one co-habiting child, ages 3 to 6 years old

  * Spouse/partner of OEF/OIF/OND veteran with at least one co-habiting child, ages 3 to 6 years old, can only participate if Veteran is participating
  * Co-habiting child (3 to 6 years) of OEF/OIF/OND veteran
  * Signed informed consents
  * Access to computer with webcam and internet access

Exclusion Criteria:

* • Does not meet the inclusion criteria

  * Either parent does not want the child to participate
  * Participated in FOCUS-EC while on active duty
  * Active psychosis/mania (as assessed by staff)
  * Significant child developmental delays (as assessed by staff)

Families excluded from the study will be provided with a list of online resources.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2014-04-03 (Actual); Primary Completion 2017-01-18 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Eyberg Child Behavior Inventory (ECBI) from baseline to 12months | Baseline and 12months
  The Eyberg Child Behavior Inventory (ECBI) will be used to obtain the frequency of problem behaviors (Intensity subscale) and whether or not the behavior is problematic for the parent (Problem subscale). The ECBI has demonstrated strong reliability, including internal consistency (.88-.95), inter-rater reliability (.79-.86), and test-retest reliability (.86-.88). It also has appropriate criterion-related validity. Both of the ECBI subscales are highly correlated with CBCL Externalizing Behavior.
Change in Strengths and Difficulties SDQ from baseline to 12 months | Baseline and 12months
  The Strengths and Difficulties Questionnaire (SDQ) is a brief emotional and behavioral screening questionnaire for children and young people. The SDQ consists of 25 items equally divided across five scales measuring emotional symptoms, conduct problems, hyperactivity-inattention, peer problems, and prosocial behavior.
Change in Spence Child Anxiety Scale-Preschool Version (SCAS) from baseline to 12 months | Baseline and 12months
  The Spence Child Anxiety Scale-Preschool Version (SCAS) Separation Anxiety, General Anxiety, and Fear of Physical Harm subscales will be used to assess child anxiety. The SCAS shows high internal consistency and test-retest reliability and was acceptable in a community sample. Positive mood, negative mood and compliance will be coded from videotaped PCI tasks; anger and compliance will be coded from the videotaped WFI tasks.
Change in Brief Symptom Inventory (BSI-18) from baseline to 12 months | Baseline and 12 months
  Parental psychological distress will be measured using the Brief Symptom Inventory. The BSI-18 measures somatization, depression, and anxiety as well as the global severity index (GSI), including all 18 items. Anxiety and depression scores were calculated by averaging the six items pertaining to each subscale (Cronbach's α = 0.88, 0.89, respectively). Scores were calculated when no more than two items were missing per subscale.
Change in Patient Health Questionnaire (PHQ9) from baseline to 12 months | Baseline and 12 months
  The PHQ-9 is the nine item depression scale of the Patient Health Questionnaire. There are two components of the PHQ-9: to assess symptoms and functional impairment to make a tentative depression diagnosis, and to derive a severity score to help select and monitor treatment. Reliability and validity of the PHQ-9 have indicated it has sound psychometric properties. Internal consistency of the PHQ-9 has been shown to be high.
Change in Parenting Stress Index (PSI-SF) from baseline to 12 months | Baseline and 12months
  Parenting stress was assessed using the 36-item Parenting Stress Index- Short Form (PSI-SF). The PSI-SF consists of three subscales: Parental Distress, Parent-Child Dysfuncitonal Interaciton (PC-DysFx), and Difficult Child. The Parental Distress subscale examines the degree of distress parents are experiencing in their parental role and was considered as a measure of parent psychological health (α = 0.89).
Change in Posttraumatic Diagnostic Scale (PDS) from baseline to 6 months | Baseline and 6 months
  Parent PTSD symptoms were assessed using the four-part Posttraumatic Diagnostic Scale (PDS). This study used the 17-item symptom severity section. Re-experiencing and Arousal scores were calculated by summing the five items pertaining to each subscale, and Avoidance scores by summing the seven items pertaining to the subscale (Cronbach's α = 0.94, 0.92, and 0.92, respectively). Total scores were calculated by summing all17 items (Cronbach's α = 0.96). PDS has high internal consistency and test-retest reliability.
Change in Parental Behavior with Preschooler Q-Sort from baseline to 12 months | Baseline and 12months
  Parents' perceptions of their sensitive parenting behaviors were assessed using nine items from the Parental Behavior with Preschooler Q-Sort, which were adapted as self-report questionnaire items (PBP-Sensitivity); the self-report items have shown predictive validity for a variety of child and parent characteristics.
Change in Parent Child Interaction (PCI)/NICHD Qualitative Rating from baseline to 12 months | Baseline and 12 months
  Each parent will also participate in a 15 minute videotaped parent-child interaction task based on the NICHD Study of Early Child Care "Three Bag" semi-structured free play procedure. Mothers and fathers will be provided with three different but comparable sets of developmentally appropriate toys, and instructed to play with the toys in a specified order. Qualitative ratings developed for the NICHD Study of Early Child Care will be used to assess parent behavior (sensitivity/supportive presence, intrusiveness, detachment/disengagement, positive regard, and negative regard) Two research assistants will be trained to reliability to code the videotaped parent-child interactions. Dr. Paley has used this coding system in her previous and current research. Approximately 20% of the interactions will be double-coded to assess inter-rater reliability. Coders will be blind to treatment condition.
Change in WFI- Whole Family Interaction/Young Family Interaction Coding System (YFICS) from baseline to 12 months. | Baseline and 12 months
  The WFI task will be used to assess family positive affect, negative affect, detachment, intrusiveness, and alliances. Families will be videotaped during a 15-minute play task in which they are asked to build something together with Duplos®. Ratings of the family interaction task will be made from videotapes using the Young Family Interaction Coding System (YFICS). The WFI has been predicted by parental attachment classifications and marital interactions and adequate reliability has been established for the YFICS. Coding will focus on the quality of interactions among all family members, rather than on interactions within any particular dyad.

SECONDARY OUTCOMES:
Change from baseline to 12 months on Coping Self Efficacy (CSE) measure | Baseline and 12 months
  The Coping Self Efficacy Scale (CSE) is a 26 item assessment that provides a measure of a person's perceived ability to cope effectively with life challenges and a way to assess changes over time. An overall CSES score is created by summing the item ratings (α = .95; scale mean = 137.4, SD = 45.6).
Change from baseline to 12 months on Home Observation for Measurement of the Environment Early Childhood Version (HOME) | Baseline and 12 months
  Home Observation for Measurement of the Environment Early Childhood Version (HOME) will be used to measure both the physical environment of the home, as well as interactions that take place there. The HOME is an interviewer rated measure based on a home visit with the child and caregiver. The Early Childhood version has eight subscales including Acceptance of Child, Learning Materials, Parental Responsivity, Physical Environment, Variety in Experience, Language Stimulation, Learning Stimulation, and Modeling of Social Maturity. The ratings are based on observation and semi-structured questions asked of the parents. Alpha coefficients for internal consistency range from .44 to .89.
Change from baseline to 12 months on Ages and Stages Questionnaire: Social Emotional (ASQ:SE) | Baseline and 12months
  Children's social-emotional competence and problem behavior will be assessed using the Ages and Stages Questionnaire: Social Emotional (ASQ:SE). The ASQ:SE is comprised of seven scales, including Self-Regulation, Compliance, Communication, Adaptive Functioning, Autonomy, Affect, and Interaction with People. The ASQ:SE has been found to have acceptable test-retest reliability,good internal consistency, and good sensitivity and specificity in identifying children at risk for social-emotional problems.
Change from baseline to 12 months on Coparenting Questionnaire | Baseline and 12 months
  The Coparenting Questionnaire will be used to assess parents' perceptions of cooperation, conflict, and triangulation among coparents. Cronbach alphas range from .69 to .87 for internal consistency.
Change from baseline to 12 months on McMaster Family Assessment Device (FAD) | Baseline and 12months
  Family Environment: Family functioning will be assessed by the McMaster Family Assessment Device (FAD). FAD includes seven subscales: Problem Solving, Communication, Roles, Affective Responsiveness, Affective Involvement, Behavior Control, and General Functioning. Home Observation for Measurement of the Environment Early Childhood Version (HOME) used to measure the physical environment of the home, as well as interactions that take place there.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Lester, MD, Principal Investigator — University of California, Los Angeles, Semel Institute; Catherine Mogil, PsyD, Study Director — University of California, Los Angeles, Semel Institute

IPD SHARING:
Plan to Share IPD: No